CLINICAL TRIAL: NCT01040507
Title: Very Long Term Results After Laparoscopic Retrocolic Antegastric Gastric Bypass
Acronym: >10yrsRYGB
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD; FACS; FASMBS; Professor of Surgery, University of California San Francisco, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2009023; U1111-1113-0364 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-23; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-08

CONDITIONS: Clinically Severe Obesity
Keywords: severe obesity; morbid obesity; gastric bypass; efficacy of gastric bypass
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- primary laparoscopic gastric bypass

SUMMARY:
The main aim of this study is to analyze and report the very long-term outcomes after primary laparoscopic proximal Roux-en-Y gastric bypass surgery for clinically severe obesity.

DETAILED DESCRIPTION:
There is lack of very-long term outcomes after bariatric surgery; A few series have been reported. However, most of them analyze medium-term outcomes. For RYGB, there are just two retrospective cohort studies reporting very long-term outcomes. Both studies have an open approach and a proximal Roux-en-Y configuration with different pouch orientation and size. MacLean´s series, with a better follow-up rate (83.4%), had a 67.6%EWL at a mean of 11.4 years; Failure rates were 20 and 35% for the morbidly obese and super obese, respectively. We will analyze our own series with a laparoscopic approach, vertically, lesser-curve base < 10-15ml pouch and proximal Roux limb. The main end-points for our study are 1) Morbidity including status of specific biochemical markers & Mortality, 2) Weight loss expressed as BMI or %EWL, 3) Trends in major comorbidities and 4) Assessment of Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* patients who met NIH criteria for recommendation of a bariatric procedure with a combination of the following characteristics

  * status post primary laparoscopic proximal RYGB surgery with or without subsequent open or laparoscopic revisions or re-operations
  * follow up > 10.0 years (Very long term outcome)

Exclusion Criteria:

* patients who had a previous gastric or bariatric procedure
* patients who underwent primary laparoscopic RYGB somewhere else by other surgical group
* missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had clinically severe obesity and underwent a primary laparoscopic Roux-en-Y Gastric Bypass more than years ago were identified form a prospectively maintained database at UCSF Fresno / ALSA med group, Inc Minimally Invasive Surgery Program.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Weight loss expressed as Body Mass Index and Percentage excess weight loss | throughout follow-up
Comorbidity status | throughout follow-up
Health-related Quality of Life (HR-QoL) | at last follow-up
Subjective satisfaction | at the last follow-up
Morbidity and mortality | throughout follow-up

SECONDARY OUTCOMES:
Nutritional and metabolic status | throughout follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Department of Surgery, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] www.asbs.org/htm/Private/resolution.html. American Society of Metabolic and Bariatric Surgeons.
- [Background] O'Brien PE, McPhail T, Chaston TB, Dixon JB. Systematic review of medium-term weight loss after bariatric operations. Obes Surg. 2006 Aug;16(8):1032-40. doi: 10.1381/096089206778026316. PMID 16901357
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Christou NV, Look D, Maclean LD. Weight gain after short- and long-limb gastric bypass in patients followed for longer than 10 years. Ann Surg. 2006 Nov;244(5):734-40. doi: 10.1097/01.sla.0000217592.04061.d5. PMID 17060766
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery